CLINICAL TRIAL: NCT05904314
Title: The Effect Of Simulation Teaching Method On Students' Knowledge, Satisfaction, And Self-Efficacy İn Electronic Fetal Monitoring Follow Up And Management
Brief Title: Evaluation of the Effectiveness of Teaching Method With Simulation in Electronic Fetal Monitoring Management
Acronym: EFM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IGULER
Record Dates: First submitted 2023-04-17; First posted 2023-06-15 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2024-06

CONDITIONS: Cardiotocography; Electronic Fetal Monitoring; High Fidelity Simulation Training
Keywords: Electro fetal monitor; high-fidelity simulation; satisfaction; self-confidence
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: 68 participants, control group theory training experimental group Electronic fetal monitor management simulation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Investigation of the effectiveness of scenario-based standardized patient simulation training and electronic fetal monitor management of midwifery students
  Interventions: Behavioral: Simulation training in electronic fetal monitor management
- Control Group (No Intervention): Behavioral: Examining the effectiveness of electronic fetal monitor management of midwifery students with theory training

INTERVENTIONS:
Behavioral: Simulation training in electronic fetal monitor management — Simulation training in electronic fetal monitor management
  Arms: Experimental Group

SUMMARY:
Electro fetal monitor monitoring in the antepartum and intrapartum periods is one of the most important responsibilities of midwives, who have important roles and responsibilities in maintaining and managing the health of women and newborns before, during and after delivery. Although midwives receive training on EFM monitoring with classical methods before graduation, they may experience problems in EFM monitoring in the clinical field after graduation. For this reason, midwife students should have the knowledge, skills and self-efficacy about a good level of EFM monitoring during their undergraduate education. In recent years, simulation-based education in the field of health has increased rapidly. This method creates an opportunity for health professionals, students, patient assessment, interaction and holistic care without compromising patient safety, and develops participants' critical thinking, clinical decision making and problem solving skills.

In this context, it is very important to evaluate the EFM trace in the antepartum and intrapartum periods, to determine the possible risks, to plan, implement and evaluate the interventions, to provide the emergency crisis management in a short time without affecting the fetal health, and to increase the self-confidence of the midwives.

The research was planned quantitatively in the form of randomized control-intervention of the scenario-based realistic simulation method, to increase the satisfaction and self-confidence levels of midwifery students in learning, to evaluate the simulation design and educational effectiveness, in EFM management. The research will facilitate midwifery students to intervene with the patient in a shorter time, with confidence and with sufficient clinical skills, and patient safety will be increased. It will also allow for the reduction of erroneous clinical practices and malpractices.

This research aims to evaluate the effect of high-fidelity simulation teaching method on knowledge, satisfaction and self-efficacy of midwifery students in EFM follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the research,
* Being a midwifery second year student and taking the "Risky pregnancy" course,
* Attending training with simulation for the first time

Exclusion Criteria:

* Incomplete filling of data collection forms,
* Not participating in all applications of simulation teaching,
* Desire to leave the research.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2025-04-10 (Estimated)

PRIMARY OUTCOMES:
information evaluation form | immediately before simulation
  The information evaluation form is in a multiple-choice format consisting of 50 questions by scanning the literature by the researchers. Each question is worth 2 points
information evaluation form | 5 weeks after the first simulation application
  The information evaluation form is in a multiple-choice format consisting of 50 questions by scanning the literature by the researchers. Each question is worth 2 points
Student Satisfaction and Self-Confidence Scale in Learning | immediately after the first simulation application
  The scale is a 13-item measurement tool designed to measure student satisfaction with simulation and self-confidence during practices. It is a 5-point Likert type and is scored as strongly disagree 1, disagree 2, undecided 3, agree 4, strongly agree 5.
Student Satisfaction and Self-Confidence Scale in Learning | immediately after the second simulation application
  The scale is a 13-item measurement tool designed to measure student satisfaction with simulation and self-confidence during practices. It is a 5-point Likert type and is scored as strongly disagree 1, disagree 2, undecided 3, agree 4, strongly agree 5.
Self-efficacy scale in monitoring and management of electronic fetal monitoring | immediately after the second simulation application
  It has been determined that the 32-item scale .Electro Fetal Monitor Monitoring Scale can be used as a valid and reliable scale in health professionals. Minimum 0, maximum 32. As the score increases, it is determined that the self-efficacy is higher.

SECONDARY OUTCOMES:
Simulation Design Scale | immediately after the first simulation application
  The simulation method applied and designed to the intervention group is used in the evaluation of the participants. The simulation design scale consists of 20 items in total. Evaluation of the scale is done in two stages. In the first stage, in order to evaluate whether the items used in the simulation method were given in the best way for the participant, they were expressed as strongly disagree, disagree, undecided, agree, strongly agree. In the second stage, there are statements that will determine the level of importance of the scale items for the participant, not important, partially important, undecided, important, very important. In the evaluation phase, the scale score is calculated by dividing the total and the total of the sub-dimensions by the number of items.
Simulation Design Scale | immediately after the second simulation application
  The simulation method applied and designed to the intervention group is used in the evaluation of the participants. The simulation design scale consists of 20 items in total. Evaluation of the scale is done in two stages. In the first stage, in order to evaluate whether the items used in the simulation method were given in the best way for the participant, they were expressed as strongly disagree, disagree, undecided, agree, strongly agree. In the second stage, there are statements that will determine the level of importance of the scale items for the participant, not important, partially important, undecided, important, very important. In the evaluation phase, the scale score is calculated by dividing the total and the total of the sub-dimensions by the number of items.
Self-efficacy scale in monitoring and management of electronic fetal monitoring | immediately after the first simulation application
  It has been determined that the 32-item scale. Electro Fetal Monitor Monitoring Scale can be used as a valid and reliable scale in health professionals. Minimum 0, maximum 32. As the score increases, it is determined that the self-efficacy is higher.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Iffet Güler Kaya, Fatih, Istanbul
  - Neriman, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
This research aims to evaluate the effect of high-fidelity simulation teaching method on knowledge, satisfaction and self-efficacy of midwifery students in EFM follow-up.
Supporting Information: Study Protocol
Time Frame: Can be used for a long time
Access Criteria: Undecided